CLINICAL TRIAL: NCT03813303
Title: Comparison of Post Anesthetic Recovery Time in Sedated Patients for Colonoscopy: Midazolam and Propofol or Fentanyl and Propofol.
Brief Title: Comparison of Post Anesthetic Recovery Time in Sedated Patients for Colonoscopy
Acronym: CPART
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Renato Santiago Gomez, Clinical Professor, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CAAE56538616230015121
Record Dates: First submitted 2018-12-27; First posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Colonoscopy; Anesthesia
Keywords: Colonoscopy; Anesthesia; Fentanyl; Midazolam; Propofol
MeSH Terms: interventions — Midazolam; Fentanyl; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Midazolam group (Active Comparator): Midazolam and Propofol administered for sedation in colonoscopy elective patients by anesthesiologist . Complications and procedure and recovery times were recorded for comparison with the Fentanyl group.
  Interventions: Drug: Midazolam; Drug: Propofol
- Fentanyl group (Active Comparator): Fentanyl and Propofol administered for sedation in colonoscopy elective patients by anesthesiologist .Complications and procedure and recovery times have were recorded for comparison with the Midazolam group.
  Interventions: Drug: Fentanyl; Drug: Propofol

INTERVENTIONS:
Drug: Midazolam — Administration of midazolam by anesthesiologist for sedation.
  Arms: Midazolam group
Drug: Fentanyl — Administration of fentanyl by anesthesiologist for sedation.
  Arms: Fentanyl group
Drug: Propofol — Administration of propofol by anesthesiologist for sedation.

SUMMARY:
Colonoscopy is an important diagnostic and therapeutic tool in colon disorders. Different drugs and levels of sedation can be used in its accomplishment. There is no consensus on which is the ideal. The aim of this study was to compare the post anesthetic recovery time between patients deeply sedated with midazolam and propofol or fentanyl and propofol. 50 American Society of Anesthesiologist physical state (ASA) I and II candidates elective colonoscopy at Luxembourg Hospital were divided into two groups A) midazolam and propofol or B) fentanyl and propofol. Time of examination, post anesthetic recovery and discharge at home, intercurrence and propofol consumption were compared.

DETAILED DESCRIPTION:
A prospective, randomized, double-blind study conducted in the complementary examination department of the Luxembourg Hospital, approved by the ethics and research committee of the Luxembourg Hospital / Mário Penna Foundation (CAAE: 56538616.2.3001.5121). The sample size was calculated in 21 participants for each group, based on a previous study, considering a standard deviation of 7.5, to detect a difference of 7.5 minutes, with a power of 90% and significance level of 5% . To cover possible losses, two groups were set up with 25 participants: midazolam and propofol, B fentanyl and propofol. Patients were invited to participate in physical status ASA I and II candidates for elective colonoscopy.

The randomization was done through the distribution of numbers generated by the site www.random.org in two groups A and B, with a sweeping draw. All participants signed a free and informed consent form. The syringes were previously prepared by the anesthesiology resident with 3mg midazolam or 50 mcg fentanyl and double distilled water to make up to 5ml volume. Patients received standard and oxygen monitoring by nasal catheter at 4 liters / minute. The anesthesiologist in charge administered a syringe delivered by the resident according to the randomization, without knowing which solution was followed, followed by 50 mg of propofol in increments of 20 mg until reaching the Ramsay stage 4 of sedation and then the physician endoscopist was authorized to introduce the colonoscope. The patient was maintained in this sedation plan until the device was withdrawn through further 20 mg increments of propofol administered according to the subjective evaluation of the anesthesiologist. Episodes of patient awakening, movement, oxygen saturation (SpO2) drop below 90%, and need for ventilatory assistance were noted if they occurred. The time between the introduction of the endoscope and its withdrawal was defined as the examination time.Then, the patient was refered to the post-anaesthesia care unit 1(PACU 1) where remained monitorized and supervised by a nurse technique and a doctor from anestehsiology team until reached the Aldrete Recovery Scale nine score. Reaching this criterion, the patient was referred to post-anaesthesia care unit 2 (PACU 2) where he remained seated, without monitoring and supplemental oxygen until he was able to walk,and drink water. Then he was discharged from the hospital. This time was noted by another nursing technique: SRPA 2 Time. Quantitative variables were submitted to the Shapiro-Wilk normality test, which is more suitable for small samples. Data that presented normal distribution (parametric data) were submitted to Student's t-Test. Non-parametric data were analyzed according to the Wilcoxon Test. The Pearson Correlation Tests (parametric data) and Spearman (nonparametric data) were used to evaluate the existence of a relationship (positive or negative) between two variables. In all tests, the obtained differences were considered statistically significant when the value of p was less than 0.05 (p <0.05). The analyzes were performed using GraphpadPrism®, version 5.0 for Windows.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II physical status patients scheduled for elective colonoscopy.

Exclusion Criteria:

* BMI less than 17 or over 30
* allergy to any medication used,
* cognitive difficulty,
* psychiatric disorder,
* hospitalization,
* chronic use of opioids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2018-06-25 (Actual)

PRIMARY OUTCOMES:
Recovery time | An average of two hours after the termination of the procedure.
  The main objective was to compare post-anesthetic recovery times, defined as a score greater than or equal to 9 on the Aldrete scale, in patients submitted to two sedation regimens: midazolam with propofol or fentanyl with propofol. Aldrete scale is a post anesthesic recovery scale that ranges from 0 to 10, meaning complete recovery in values above nine.

CONTACTS AND LOCATIONS:
Overall Officials: Renato Gomez, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Luxemburgo Hospital, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No